CLINICAL TRIAL: NCT03531723
Title: Brain Ultrasound in the Weaning of External Ventricular Leads
Acronym: ECHO-SD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/18/0178; 2018-A01219-46 (Other: ID-RCB)
Record Dates: First submitted 2018-05-09; First posted 2018-05-22 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Hydrocephalus; Intracranial Hypertension
Keywords: external ventricular derivation
MeSH Terms: conditions — Hydrocephalus; Intracranial Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Measuring the size of the 3rd ventricle by ultrasound — The surveillance of the clamping test is essentially clinical. No cerebral imaging is performed systematically in our service protocol.The study consisted of including ultrasound measurements during the usual weaning protocol of the service.All patients receiving a SEV withdrawal test will be included. Inclusion begins when the clinician in charge of the patient initiates the withdrawal test. The measurements will be performed blindly by a trained physician who does not participate in the patient's care. Four measurements will be made, with recording of ultrasound loops

SUMMARY:
External Ventricular Deviation (EDV) is a medical device that provides transient and controlled external drainage of cerebrospinal fluid (CSF). This device can also monitor intracranial pressure (ICP). SEV is an emergency measure indicated for acute hydrocephalus and / or intracranial hypertension (HTIC). Weaning from a DVE should be considered as soon as possible from the moment the patient's clinical condition allows it. There is no consensus on how to wean SEVs.

The main objective of this study is to evaluate inter and intraobserver reproducibility of the measurement of the 3rd ventricle size by ultrasound in patients receiving a DVE withdrawal test.

DETAILED DESCRIPTION:
Ultrasound assessment of the ventricular system, including the size of the 3rd ventricle, can be used in severe traumatic brain injury. Ultrasound measurement of the size of the 3rd ventricle is used as a marker to monitor cerebral atrophy in neurodegenerative diseases such as multiple sclerosis (MS). There is good correlation between brain ultrasound and MRI and CT brain imaging to assess the size of the 3rd ventricle. Ultrasound measurement of the size of the 3rd ventricle has never been evaluated in weaning external ventricular leads.

Measuring the size of the 3rd ventricle by ultrasound could be an interesting monitoring technique during a SEV withdrawal trial to predict success or failure.

Weaning is usually based on a clamp test with more or less paraclinical clinical monitoring. The recurrence of hydrocephalus and / or HTIC defines a withdrawal failure of the drainage device.

The size of the 3rd ventricle evaluated by cerebral CT in a clamp test is found as a predictor of weaning failure of a DVE.

ELIGIBILITY:
Inclusion Criteria:

* Patient benefiting from a DVE, whatever the indication
* Hospitalized in the neurosurgical resuscitation and neurosurgical intensive care units of Toulouse University Hospital
* First DVE withdrawal test initiated by the doctor in charge of the patient
* Major patient
* Affiliated person or beneficiary of a social security scheme.
* Expression of non-opposition by the participant or his / her confidant and the investigator (at the latest on the day of inclusion and before any examination required by the research).

Exclusion Criteria:

* Absence of cerebral acoustic window
* Patient with a ventriculoperitoneal (DVP) diversion before the DVE.
* Antecedent surgery in the cerebral ventricular system.
* Pregnant and lactating woman
* Person under safeguard of justice
* Nosocomial neuro-meningeal infection on untreated or treatment-emergent DVE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years-old, receiving a DVE withdrawal test and hospitalized in the neurosurgical resuscitation and neurosurgical intensive care units of Toulouse University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-07-12 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Inter individual reproducibility of ultrasound measurement of the size of the 3rd ventricle | 3 weeks
  Inter individual reproducibility of ultrasound measurement of the size of the 3rd ventricle at different study times The inter-individual reproducibility will be evaluated at each time by the analysis of a loop by 3 independent and blind operators.
  The analysis of all ultrasound loop recordings will be performed at the end of the participation of the last included patient. The recordings of the ultrasound loops will be coded and presented in a random and different order to each operator.
Intra individual reproducibility of ultrasound measurement of the size of the 3rd ventricle | 3 weeks
  Intra individual reproducibility of ultrasound measurement of the size of the 3rd ventricle at different study times The intra-individual reproducibility will be evaluated at each time by the acquisition of 3 ultrasound loops analyzed by the same operator.
  The analysis of all ultrasound loop recordings will be performed at the end of the participation of the last included patient. The recordings of the ultrasound loops will be coded and presented in a random and different order to each operator.

SECONDARY OUTCOMES:
Measurement of the evolution of the size of the 3rd ventricle (intra individual) | 3 weeks
  Intra individual reproducibility of the ultrasound measurement of the evolution of the size of the 3rd ventricle
Measurement of the evolution of the size of the 3rd ventricle (inter individual) | 3 weeks
  Inter individual reproducibility of the ultrasound measurement of the evolution of the size of the 3rd ventricle
Successful completion of the DVE withdrawal test | 3 weeks
  Successful completion of the DVE withdrawal test, defined by the absence of the need to decline or rest a DVE at 3 weeks.
Failure of the weaning test | 3 weeks
  Failure of the weaning test defined by the need to decline or rest a DVE at 3 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Timothée ABAZIOU, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No